CLINICAL TRIAL: NCT05253417
Title: The CANabidiol Use for RElief of Short Term Insomnia (CAN-REST). A Randomised, Double-Blind, Placebo-Controlled Clinical Study
Brief Title: The CANabidiol Use for RElief of Short Term Insomnia
Acronym: CANREST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bod Australia (Industry)
Collaborators: Woolcock Institute of Medical Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BOD202101
Record Dates: First submitted 2021-12-20; First posted 2022-02-23 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Sleep Disturbance; Insomnia; Insomnia Type; Sleep Disorder; Insomnia, Transient; Insomnia Due to Anxiety and Fear; Insomnia Due to Other Mental Disorder
Keywords: Insomnia; sleep; fatigue; cannabidiol; CBD; mental health; anxiety
MeSH Terms: conditions — Parasomnias; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Fatigue; Psychological Well-Being; Anxiety Disorders | interventions — Cannabidiol; Capsules

STUDY DESIGN:
Intervention Model Description: Randomised, placebo-controlled, double-blind, parallel trial
Who Masked: Participant, Investigator
Masking Description: Double-blind: Study staff (including the study investigators, the clinical trials coordinator and the study medical officer) and the participants will be blinded. Blinding will be maintained by the use of identical containers and labels except for the patient identification code and unique batch number.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 50 mg CBD (Experimental): 50 mg CBD to be administered as a single oral dose. Each capsule contains 25 mg CBD. Two capsules to be taken (plus two placebo capsules)
  Interventions: Drug: 50 mg Cannabidiol (CBD); Drug: Placebo; Drug: 100 mg Cannabidiol (CBD)
- 100 mg CBD (Experimental): 100 mg CBD to be administered as a single oral dose. Each capsule contains 25 mg CBD. Four capsules to be taken.
  Interventions: Drug: 50 mg Cannabidiol (CBD); Drug: 100 mg Cannabidiol (CBD)
- Placebo (Placebo Comparator): Placebo capsules contain no CBD. Four capsules to be taken as a single oral dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 50 mg Cannabidiol (CBD) — For the study arm, '50 mg CBD' participants take two (2) CBD capsules and two (2) placebo capsules.
  Other Names: BodECS BioAbsorb(TM) capsule
  Arms: 100 mg CBD; 50 mg CBD
Drug: Placebo — Participants take four (4) placebo capsules.
  Arms: 50 mg CBD; Placebo
Drug: 100 mg Cannabidiol (CBD) — For the study arm, '100 mg CBD' participants take four (4) CBD capsules.
  Other Names: BodECS BioAbsorb(TM) capsule
  Arms: 100 mg CBD; 50 mg CBD

SUMMARY:
This study aims to investigate the effect of 50 mg and 100 mg per day oral CBD product versus a placebo over 8 weeks on insomnia severity in adults aged 18-65 years old with insomnia symptoms.

DETAILED DESCRIPTION:
This is a double-blind, randomised, parallel-group, placebo-controlled study of 8 weeks of oral CBD at 50 or 100 mg per day versus placebo in 198 participants with insomnia symptoms as classified by an Insomnia Severity Index (ISI) score of 8-21. Participants will be recruited voluntarily and are able to withdraw at any time. The study will be conducted online with telehealth consults where required.

ELIGIBILITY:
Inclusion Criteria:

1. Male and females aged 18-65 years old, inclusive.
2. Females must be non-pregnant, non-lactating.
3. Proficient in English and have internet access and a mobile phone.
4. Insomnia symptoms as classified by an Insomnia Severity Index (ISI) score of 8 - 21 and have experienced these symptoms over the past month at pre-screening.
5. Stated willingness to comply with all study procedures and availability for the duration of the study.
6. Provision of signed and dated informed consent form.
7. All male and females of childbearing potential must agree to use two forms of effective contraception from the time of signing informed consent until 30 days after study completion.

Exclusion Criteria:

1. Serious medical and/or psychiatric illnesses/disorders that will require treatment during the trial period.
2. The use of any drug known to affect sleep during the study one week prior the randomization, including:

   1. Sedatives (benzodiazepines, Z drugs, agomelatine, suvorexant, sodium oxybate, sedating antidepressants, sedating antihistamines, antipsychotics, melatonin, valerian).
   2. Opioids (e.g. morphine, codeine, oxycodone, methadone, buprenorphine, fentanyl, tramadol, tapentadol, hydromorphone).
   3. Stimulants (e.g. methylphenidate, dexamphetamine, modafinil, phentermine).
3. Excessive caffeine use (defined as > 600mg caffeine or approximately 6 cups of caffeinated beverages a day) that, in the opinion of the medical doctor, contributes to the participant's insomnia.
4. Excessive alcohol use (defined as per NHMRC guideline, i.e. no more than four standard drinks per day on average for men, and for women, no more than two).
5. The use of cannabinoids or a cannabinoid-based medicine within 3 months prior to study Day 1 and unwillingness to abstain from recreational drug use during the study period.
6. Cannabis dependence or any other drug or alcohol dependence within the past two years.
7. Positive urine drug screen (e.g., amphetamines type substances, benzodiazepines, cannabinoids, cocaine, and opiates) at screening or Day -1 or a history of drug abuse within the past 2 years.
8. Known hypersensitivity to cannabis-based products or any of the excipients in the study drug.
9. Use of any investigational drug or involvement in another clinical trial within 30 days of screening day.
10. Use of anti-coagulant drugs such as warfarin or those known to be metabolised by CYP450 enzymes.
11. Current or ongoing treatments for insomnia (e.g. cognitive-behavioural therapy (CBT) and CNS-active drugs).
12. Obstructive sleep apnoea determined by the MAPI questionnaire or other self-reported sleep disorders.
13. Medical conditions that result in frequent sleep disturbance (e.g. nocturia).
14. History of attempted suicide in the past 12 months.
15. Clinically significant hepatic abnormalities determined by the screening blood test.
16. Shift work, jet lag or trans-meridian travel (two time zones) in the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
To investigate the effect of the administration of a 50mg and 100mg per day oral CBD product versus placebo over 8 weeks on insomnia severity index scores | Baseline (week 0), week 4, week 8
  Insomnia Severity Index (ISI): A 7-item tool measuring the nature, severity, and impact of insomnia over the past 2 weeks. Each item uses a 5-point Likert scale to capture a rating (0 = no problem; 4 = very severe problem) which add up to: no insomnia (0 - 7); sub-threshold insomnia (8 - 14); moderate insomnia (15 - 21); and severe insomnia (22 - 28).

SECONDARY OUTCOMES:
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on wake after sleep onset (WASO) as assessed by actigraphy. | Baseline (week 0), week 8
  WASO is a parameter that examines the total amount of minutes awake after the first sleep epoch is achieved. Therefore, as the WASO increases, sleep efficiency decreases.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Anxiety as assessed by the DASS-21 questionnaire. | Baseline (week 0), Week 4, week 8
  Depression Anxiety Stress Scale-21 (DASS-21): A 21-item tool with subscales measuring the negative emotional states of depression, anxiety, and stress separately. Depression ranges from normal (0-9) to extremely severe (28+); anxiety ranges from normal (0-7) to extremely severe (20+); and stress ranges from normal (0-14) to extremely severe (34+).
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Stress as assessed by the DASS-21 questionnaire. | Baseline (week 0), Week 4, week 8
  Depression Anxiety Stress Scale-21 (DASS-21): A 21-item tool with subscales measuring the negative emotional states of depression, anxiety, and stress separately. Depression ranges from normal (0-9) to extremely severe (28+); anxiety ranges from normal (0-7) to extremely severe (20+); and stress ranges from normal (0-14) to extremely severe (34+).

OTHER OUTCOMES:
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Sleep onset latency (SOL) measured by actigraphy. | Baseline (week 0), week 8
  Sleep onset latency (SOL) is the time it takes to transition from wakefulness to non-REM sleep. On average, the SOL should take between 10-20 minutes. Short sleep latencies usually reflect increased sleepiness.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on subjective sleep as assessed by sleep diaries | Baseline (week 0), week 4, week 8
  Participants will be requested to complete a short, 5-minute online sleep diary for seven mornings to describe the previous night's sleep at baseline, week 4 and week 8.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on self-perception of improvement in sleep as assessed by a self-report questionnaire. | Baseline (week 0), week 4, week 8
  The self-report questionnaire will ask participants to rate their self-perceived improvement in sleep using a standard 10-point visual analogue scale at weeks 4 and 8
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Subjective sleep-related quality of life as assessed by the Functional Outcomes Sleep Questionnaire (FOSQ-10). | Baseline (week 0), week 4, week 8
  FOSQ-10 is a 10 items questionnaire to measure the impact of daytime sleepiness on activities of daily living. The score range is 5-20 points, with higher scores indicating better functional status.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Fatigue assessed by the Flinders Fatigue Scale; | Baseline (week 0), week 4, week 8
  The Flinders Fatigue Scale is a 7 items self-report scale which assess fatigue over the past 2 weeks. This scale provides a total fatigue score ranging from 0 to 31, with higher scores indicating greater fatigue.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Health-related quality of life (HRQoL) assessed using the EQ-5D-5L. | Baseline (week 0), week 4, week 8
  A descriptive system for health-related quality of life states in adults, consisting of five dimensions. Each of which has five severity levels that are described by statements appropriate to that dimension. Those are rated by a verbal 5-point rating scale allowing for distinction of five levels ('5L') of severity: Level 1: no problems; Level 2: slight problems; Level 3: moderate problems; Level 4: severe problems; Level 5: extreme problems per dimension and providing a 1-digit number for each dimension.
To determine the effect of 8 weeks of 50mg or 100mg of CBD on the number of participants with treatment-emergent adverse events | Week 4, Week 8, Week 12
  The safety and tolerability of the investigational product will be determined by evaluating all incidences of treatment-emergent adverse events as assessed by reported by participants or observed by the investigators or from the safety pathology tests.
To determine relationship between efficacy endpoint and systemic concentrations of CBD and its carboxy and hydroxy metabolites | Baseline (week 0), week 8
  Systemic concentrations of CBD (ng/mL), 7- hydroxycannabidiol (7-OH-CBD) (ng/mL) and 7- carboxycannabidiol (7- COOH-CBD) (ng/mL) will be analysed in plasma and urine samples collected at baseline and week 8.
To determine the effect of 8 weeks of 50mg or 100mg of CBD compared to placebo on Depression as assessed by the DASS-21 questionnaire. | Baseline (week 0), Week 4, week 8
  Depression Anxiety Stress Scale-21 (DASS-21): A 21-item tool with subscales measuring the negative emotional states of depression, anxiety, and stress separately. Depression ranges from normal (0-9) to extremely severe (28+); anxiety ranges from normal (0-7) to extremely severe (20+); and stress ranges from normal (0-14) to extremely severe (34+).

CONTACTS AND LOCATIONS:
Overall Officials: Ron Grunstein, Principal Investigator — Woolcock Institute of Medical Research
Locations (2):
- Australia (2):
  - Woolcock Institute, Glebe, New South Wales
  - Fusion Clinical Research, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No